CLINICAL TRIAL: NCT03592225
Title: Prevention At PRImary CAre Level - Increasing HPV Vaccination in Lyon.
Brief Title: Can an Educational Intervention Targeting General Practitioners Increase HPV Vaccination Coverage in AuRA_Lyon (France)
Acronym: PAPRICA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: International Agency for Research on Cancer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PP201704-07
Record Dates: First submitted 2018-04-19; First posted 2018-07-19 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Human Papillomavirus Vaccination
Keywords: General Practitioners; France; RCT; HPV vaccination

STUDY DESIGN:
Intervention Model Description: 2 groups of General practitioners are randomized to be allocated either in the intervention group or the control group
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational workshop intervention arm (Other): The group of general practitioners (GP) from Lyon (France), about 300, that will be invited to attend the 3 hours educational workshop about HPV vaccination. After the workshop, the GPs will return to their normal health care practice.
  Interventions: Behavioral: Educational workshop
- Control arm (No Intervention): The group of general practitioners (GP) from Lyon (France), about 300, that will NOT be invited to attend the 3 hours educational workshop about HPV vaccination. These GPs perform their normal health care practice.

INTERVENTIONS:
Behavioral: Educational workshop — the intervention is a 3 hours educational workshop designed to address all the potential questions that the general practitioners (GP) and their patients might have regarding HPV vaccination.
  Arms: Educational workshop intervention arm

SUMMARY:
The PAPRICA implementation trial aims to test the efficacy of an educational intervention about HPV vaccination and targeting general practitioners in Lyon

DETAILED DESCRIPTION:
The PAPRICA study aims to test if an intervention directed to General Practitioners (GP) to train them in methods for recommending HPV vaccine with greater confidence and efficiency is effective to increase HPV vaccination coverage in France. As each health professional is associated in France to a specific reference number i.e. "RPPS number", RPPS numbers for all General Practitioners (GP) from the city of Lyon will be randomly allocated either to the intervention arm or to the control arm to ensure that each arm contains 50% of the total number of GPs. After allocation, GPs in the allocation arm will be identified and invited to attend the intervention i.e. a 3-hour workshop at IARC in the presence of HPV vaccination specialists. The effect of the intervention on the HPV vaccination coverage in Lyon will be measured through HPV vaccines reimbursement data extracted from the Inter-Scheme National Information System within the National Health Insurance System (SNIIR-AM : Système National d'Information Inter-Régimes de l'Assurance Maladie ). Linkable data between girls and General Practitioners (GP) via RPPS numbers will allow us to allocate girls either in the intervention or the control arm. Vaccination coverage will be estimated within each of these cohorts.

ELIGIBILITY:
Inclusion Criteria:

* general practitioners (GP) from Lyon (69001-69009) from private practice

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Assessing change from baseline HPV vaccination coverage of Lyon's girls aged 11-14 obtained by the GP from the intervention arm at 18 months after the intervention (increase in number of vaccinated girls as assessed by questionnaire in the study cohort) | 18 months
  The French SNIIRAM (Système national d'information inter-régimes de l'assurance maladie) database will be used to calculate a proxy of HPV vaccination coverage. SNIIRAM contains anonymous and individualized data for all health expenditure claims in France. Data related to HPV and DTP (Diphtheria,Tetanus, Pertussis) vaccines prescribed by GP from Lyon will be extracted from SNIIRAM for girls aged 10-14. These data will be assigned either to the intervention or control arm by linkage with GP's ID DTP booster coverage, which is stable overtime and very high in France (92%), will be used as a control.

SECONDARY OUTCOMES:
Assessing change from baseline in GP's attitude and knowledge towards HPV vaccination 1 month after receiving the intervention | 1 month
  GP's attitude and knowledge towards HPV vaccination will be assessed before and 1 month after the intervention through a specific questionnaire designed to measure GP's knowledge and beliefs upon HPV vaccination.

OTHER OUTCOMES:
3. Assessing change from control group in mothers and girls' attitude and knowledge towards HPV vaccination 18 months after the intervention | 18 months
  Parents and girls whose GP are in the intervention arm will be interviewed 18 months after the intervention to assess whether or not their attitude towards HPV vaccination has changed. Parents and girls whose GP are in the control arm will be used as control.

CONTACTS AND LOCATIONS:
Overall Officials: PATRICIA VILLAIN, PhD, Principal Investigator — IARC, WHO
Locations (1):
- International Agency for Research on Cancer (IARC), Lyon, France

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication will be shared after anonymization performed by the PI
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: from March 2016 to October 2020
Access Criteria: (1)Data from RPSS and SNIIRAM databases and data originated from original data analysis: All data will be stored in encrypted and password-locked files at IARC, while transmission of information via electronic means will be performed using encrypted data files. Measures ensuring confidentiality of personel data will be used. (2) Data generated from GPs: Data collected from questionnaires and focus groups will be anonymous, aggregated and no linkage between GP's opinion and attitude about vaccination and identity will be possible. Data will be kept and used according to the Data Protection Act (DPA). The Data Protection Act (DPA) of 1978 (revised in 2004) is the main law protecting data privacy in France. Data from GPs will be stored in encrypted and password-locked files at IARC. Only anonymised data will be transferred to IARC external collaborators.